CLINICAL TRIAL: NCT04555473
Title: Translational Analysis In Longitudinal Series of Ovarian Cancer ORganoids
Acronym: TAILOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: TAILOR
Record Dates: First submitted 2020-05-25; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-04

CONDITIONS: Organoids; Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — Bioptic tissue from the tumor will be collected from PDS and NACT+IDS patients at the time of surgery. Part of the bioptic tissue will be used to obtain organoids, whereas part will be frozen for direct comparative analysis of the original tumor. Blood samples will also be collected to purify extracellular circulating RNA (cRNAs).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Tumor biopsy — Both interventions performed at baseline upon study enrolment (pre- and post-NACT for NACT+IDS patients) and at the time of recurrence.
  1. Part of each surgical specimen will be used to obtain organoids, whereas part will be frozen for direct comparative analysis of the original tumor (1-6 organoids from each patient).
  2. Blood samples will be collected to purify extracellular circulating RNA (cRNAs).
  Other Names: Blood sampling

SUMMARY:
This is a longitudinal observational phase II, single center, single arm study on the reliability of high grade serous ovarian carcinoma organoids obtained from primary debulking surgery (PDS)+adjuvant chemotherapy and neoadjuvant chemotherapy + interval debulking surgery (NACT+IDS) cases as model for the patients' response to treatments. Since organoids represent a model system comparable to patient-derived xenografts, the investigators tested the null hypothesis that the possibility of correctly identifying the drug-sensitivity could improve from 80%, as assessed by xenografts to at least 95%. The first step was planned to include 7 patients; if 5 or more patients do not respond, the trial will be terminated. If the trial goes on to the second stage, a total of 43 patients will be studied. Considering a patient dropout of approximately 10%, the study was planned to enroll at least 48 patients.

DETAILED DESCRIPTION:
In this project, the investigators propose to employ the patients-derived organoid technology to test HGSOC organoids obtained from PDS+adjuvant chemotherapy and NACT+IDS cases to predict patients' response to treatments; moreover, the investigators aim to study genomic and phenotypic evolution of HGSOC organoids from PDS+adjuvant chemotherapy and NACT+IDS patients undergoing relapse. Finally, the investigators intend to investigate splicing-targeting technologies as new potential therapeutic treatments to increase vulnerability of HGSOCs. FIGO stage IIIC or IV ovarian, fallopian tube, or primary peritoneal cancer patients will be included if disease at metastatic sites is supposed to be completely resectable and they will be triaged for staging laparoscopy to obtain histologic diagnosis and to provide the tumor load assessment through the laparoscopic score. If PDS is chosen, open cytoreduction will be performed at the same time and bioptic tissue will be collected for organoids; otherwise, women will be submitted to NACT followed by IDS and tissue for organoids will be collected from both staging LPS biopsy (pre-) and subsequent surgery (post-NACT). Part of each surgical specimen will be used to obtain organoids, whereas part will be frozen for direct comparative analysis of the original tumor. 1-6 organoids from each patient will be prepared from PDS or NACT-IDS patients (pre- and post-NACT) and blood samples will also be collected to purify extracellular circulating RNA (cRNAs).

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 75 years
2. estimated life expectancy of at least 4 weeks
3. performance status (PS) according to Eastern Cooperative Oncology Group (ECOG) < 2
4. adequate bone marrow, respiratory, hepatic, cardiologic medullary and renal function (creatinine clearance < 60 ml/min according to Cockroft formula)
5. histologic diagnose of epithelial ovarian cancer at frozen section and laparoscopic score ≥ 8 or ≤ 12 (considered HTL) with no evidence of mesenteric retraction

Exclusion Criteria:

1. Pregnancy or breast-feeding
2. History of concomitant or previous malignancy in the last 5 years

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients
Study Population: Eligible population included women with preoperative clinical, serological and radiologic suspicion of International Federation of Gynecology and Obstetrics (FIGO) stage IIIC or IV ovarian, fallopian tube, or primary peritoneal cancer, and histological confirmation of diagnosis for HGSOC. Stage IV patients were included only in case of positive pleural effusion, or any resectable disease. All women were required to sign written informed consent to enter the study.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2020-05-12 (Actual); Primary Completion 2021-11-04 (Estimated); Study Completion 2023-05-04 (Estimated)

PRIMARY OUTCOMES:
Reliability (yes/no) of HGSOC organoids obtained from PDS+adjuvant chemotherapy and NACT+IDS cases as a model for the patient's response to treatments | Up to 36 months
  Part of each surgical specimen of eligible women will be used to obtain PDOs according to established protocols (Tuveson et al.), whereas part will be frozen for direct comparative analysis of the original tumor. At first passages, organoids will be characterized for histologic and cytologic features. PDOs maintaining HGSOC features will be analysed for genomic features and splicing-sensitive transcriptomic signatures by next generation sequencing (NGS). The identified transcriptomic signatures of PDOs will be compared to those of the original tumor by quantitative real time PCR (qPCR) analysis. PDOs will then be characterized for their response to specific drugs and the response will be compared to that of the patient undergoing chemotherapy. Dichotomic variable: Yes/No

SECONDARY OUTCOMES:
The genomic and phenotypic evolution of tumor cells in HGSOC organoids from PDS+ adjuvant chemotherapy and NACT+IDS patients undergoing relapse | Up to 36 months
  At time of relapse (if any), we will repeat NGS genomic and transcriptomic analysis of chemoresistant PDOs derived from selected patients who experienced relapse and underwent secondary surgery. Bioinformatics analyses will be applied to capture changes in the mutational status and in the transcriptional/splicing signature that accompany acquisition of chemoresistance in vitro. These features will then be compared to evolution of the tumor in vivo by sequencing (mutations) and qPCR (transcriptomics) of tissue obtained during surgery. Dichotomic variable: Yes/No
Splicing dysregulation and splicing-targeting technologies as new potential therapeutic treatments to increase vulnerability of MYC-overexpressing HGSOCs | Up to 36 months
  HGSOCs often display amplification of MYC, an oncogene that dysregulates the splicing program. We will test if HGSOC PDOs are sensitive to splicing-targeting drugs (E7107, THZ531, PRMT5 inhibitor) administered either alone or in combination with chemotherapy. THZ531 renders BRCA1/2 proficient HGSOC cell lines sensitive to PARPi. We will extend this study to PDOs and analyze their sensitivity to splicing-targeting drugs during their evolution in vitro. Changes in splicing signatures will be evaluated and correlated with the response to combined treatments, to determine their potential as biomarkers. We will also silence splicing factors deregulated in HGSOCs by RNA interference to determine their impact on PDO response to chemotherapy in terms of survival, expansion potential and transcriptomic signatures. Dichotomic variable: Yes/No

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Vizzielli, PhD, Principal Investigator — Fondazione Policlinico "A. Gemelli" IRCCS; Giovanni Scambia, Professor, Study Director — Fondazione Policlinico "A. Gemelli" IRCCS - Università Cattolica del Sacro cuore; Claudio Sette, Professor, Study Director — Catholic University of the Sacred Heart; Camilla Nero, PhD, Study Chair — Fondazione Policlinico "A. Gemelli" IRCCS; Eleonari Cesari, PhD, Study Chair — Catholic University of the Sacred Heart; Salvatore Gueli Alletti, MD, Study Chair — Fondazione Policlinico "A. Gemelli" IRCCS; Marco Pieraccioli, PhD, Study Chair — Catholic University of the Sacred Heart; Carolina Bottoni, MD, Study Chair — Fondazione Policlinico "A. Gemelli" IRCCS; Carmine Conte, MD, Study Chair — Fondazione Policlinico "A. Gemelli" IRCCS; Matteo Loverro, MD, Study Chair — Catholic University of the Sacred Heart; Anna Fagotti, Professor, Study Chair — Catholic University of the Sacred Heart
Locations (1):
- Fondazione Policlinico Universitario "A. Gemelli" IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fagotti A, Ferrandina G, Vizzielli G, Fanfani F, Gallotta V, Chiantera V, Costantini B, Margariti PA, Gueli Alletti S, Cosentino F, Tortorella L, Scambia G. Phase III randomised clinical trial comparing primary surgery versus neoadjuvant chemotherapy in advanced epithelial ovarian cancer with high tumour load (SCORPION trial): Final analysis of peri-operative outcome. Eur J Cancer. 2016 May;59:22-33. doi: 10.1016/j.ejca.2016.01.017. Epub 2016 Mar 19. PMID 26998845
- [Result] Petrillo M, Zannoni GF, Beltrame L, Martinelli E, DiFeo A, Paracchini L, Craparotta I, Mannarino L, Vizzielli G, Scambia G, D'Incalci M, Romualdi C, Marchini S. Identification of high-grade serous ovarian cancer miRNA species associated with survival and drug response in patients receiving neoadjuvant chemotherapy: a retrospective longitudinal analysis using matched tumor biopsies. Ann Oncol. 2016 Apr;27(4):625-34. doi: 10.1093/annonc/mdw007. Epub 2016 Jan 17. PMID 26782955
- [Result] Vizzielli G, Costantini B, Tortorella L, Petrillo M, Fanfani F, Chiantera V, Ercoli A, Iodice R, Scambia G, Fagotti A. Influence of intraperitoneal dissemination assessed by laparoscopy on prognosis of advanced ovarian cancer: an exploratory analysis of a single-institution experience. Ann Surg Oncol. 2014 Nov;21(12):3970-7. doi: 10.1245/s10434-014-3783-6. Epub 2014 May 22. PMID 24849521
- [Result] Hill SJ, Decker B, Roberts EA, Horowitz NS, Muto MG, Worley MJ Jr, Feltmate CM, Nucci MR, Swisher EM, Nguyen H, Yang C, Morizane R, Kochupurakkal BS, Do KT, Konstantinopoulos PA, Liu JF, Bonventre JV, Matulonis UA, Shapiro GI, Berkowitz RS, Crum CP, D'Andrea AD. Prediction of DNA Repair Inhibitor Response in Short-Term Patient-Derived Ovarian Cancer Organoids. Cancer Discov. 2018 Nov;8(11):1404-1421. doi: 10.1158/2159-8290.CD-18-0474. Epub 2018 Sep 13. PMID 30213835
- [Result] Ricci F, Bizzaro F, Cesca M, Guffanti F, Ganzinelli M, Decio A, Ghilardi C, Perego P, Fruscio R, Buda A, Milani R, Ostano P, Chiorino G, Bani MR, Damia G, Giavazzi R. Patient-derived ovarian tumor xenografts recapitulate human clinicopathology and genetic alterations. Cancer Res. 2014 Dec 1;74(23):6980-90. doi: 10.1158/0008-5472.CAN-14-0274. Epub 2014 Oct 10. PMID 25304260
- [Result] Tuveson D, Clevers H. Cancer modeling meets human organoid technology. Science. 2019 Jun 7;364(6444):952-955. doi: 10.1126/science.aaw6985. PMID 31171691